CLINICAL TRIAL: NCT07035639
Title: Exploring the Role of Baduanjin on Lumbar and Hip Mobility Index in Obese People Based on Infrared Thermography and Meridian Point Specificity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chengdu Sport University (Other)
Responsible Party: Principal Investigator, Rui Li, PhD, Chengdu Sport University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018NO.03-2024NO.04
Record Dates: First submitted 2025-06-16; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2022-09

CONDITIONS: Obesity and Overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Baduanjin group (Experimental): The Baduanjin group received training guided by national-level social sports instructors certified by the Institute of Sports Medicine, General Administration of Sport of China. The intervention consisted of Baduanjin training 4 times per week for 8 consecutive weeks, with a total duration (including warm-up and breaks) of ≥30 minutes per session. The training protocol included 16 minutes of Baduanjin exercise, a 2-minute break, and an additional 16 minutes of Baduanjin exercise.
  Interventions: Behavioral: The Baduanjin intervention was designed following traditional Chinese health preservation principles and conducted under the guidance of certified instructors. The training sessions were led by nation
- The blank control group (No Intervention): The blank control group received no exercise intervention and was advised to engage in no more than 3 sessions of aerobic exercise per week during the study. Participants in the Baduanjin group were prohibited from undertaking any other form of exercise training throughout the research period.

INTERVENTIONS:
Behavioral: The Baduanjin intervention was designed following traditional Chinese health preservation principles and conducted under the guidance of certified instructors. The training sessions were led by nation — The Baduanjin group received training guided by national-level social sports instructors certified by the Institute of Sports Medicine, General Administration of Sport of China. The intervention consisted of Baduanjin training 4 times per week for 8 consecutive weeks, with a total duration (including warm-up and breaks) of ≥30 minutes per session. The training protocol included 16 minutes of Baduanjin exercise, a 2-minute break, and an additional 16 minutes of Baduanjin exercise.
  Arms: The Baduanjin group

SUMMARY:
This study aimed to explore whether Baduanjin, a traditional fitness practice, can improve waist and hip mobility in obese individuals. Based on the TCM theory that "acupoints have unique effects," researchers hypothesized that Baduanjin might regulate muscle function by stimulating key abdominal and lumbar acupoints (such as Shenque and Guanyuan), thereby enhancing body flexibility.

The study recruited 60 overweight adults (BMI >28) from Beijing and Suzhou, randomly dividing them into two groups: one practiced Baduanjin 4 times a week for 8 weeks, while the other received no additional exercise. Using an infrared thermography device (similar to a "body temperature camera"), researchers measured temperature changes at abdominal and lumbar acupoints. They also evaluated waist mobility through forward bending, backward extension, and lateral flexion tests.

After 8 weeks, the Baduanjin group showed three significant improvements compared to the control group:

Enhanced flexibility: Waist and hip range of motion increased, such as reaching further during sit-and-reach tests.

Higher acupoint temperature: Skin temperature around Shenque, Guanyuan, and other acupoints rose, possibly indicating improved local blood circulation.

Better functional scores: Scores reflecting daily activity comfort and joint health significantly improved, while the control group showed no change.

In conclusion, Baduanjin may benefit obese individuals by "activating" abdominal and lumbar acupoints to optimize muscle function and mobility. Further research is needed to validate the underlying mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* Participants with scores of 72 or above on the HEFESCM-36 scale of the China Association of Chinese Medicine, and meeting the following criteria:

Aged between 18 and 60 years; Able to independently participate in activities required for the physical study; Body mass index (BMI) >28; No musculoskeletal diseases or radiculopathy within one year prior to the trial; No receipt of physical therapy or surgical treatment within one year prior to the trial; Education level of high school or above; Proficient in using the WeChat check-in program; No mental illnesses and with normal learning and communication abilities; Agree to and voluntarily sign the informed consent form for trial participation.

Exclusion Criteria:

* Participants with confirmed specific etiologies, such as lumbar disc herniation, lumbar fracture, etc.; Individuals with 神经根 compression symptoms, such as sciatica, lumbar disc herniation, etc.; Cases with bacterial or aseptic inflammatory diseases, such as fever, rheumatoid arthritis, etc.; Subjects with other organ pathologies, such as kidney stones, typhlitis, appendicitis, etc.; Pregnant women; Individuals taking medications for mental disorders; Participants engaging in aerobic exercise >3 times/week or anaerobic exercise >4 times/week.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2023-10-25 (Actual); Primary Completion 2023-11-25 (Actual); Study Completion 2024-01-10 (Actual)

PRIMARY OUTCOMES:
Infrared Thermography | 10min
  Used for detecting human body surface temperature

CONTACTS AND LOCATIONS:
Locations (1):
- China Academy of Chinese Medical Sciences Guang'anmen Hospital, Beijin, Beijin, China

IPD SHARING:
Plan to Share IPD: No
Unpublished IPD may contain measurement errors, missing records, or supplementary data that failed ethical review, and direct sharing could lead to deviations in secondary analysis conclusions.